CLINICAL TRIAL: NCT04722991
Title: A Phase 2 Randomized, Placebo-controlled, Double-masked Proof-of-concept Study to Investigate the Efficacy and Safety of Runcaciguat (BAY 1101042) in Patients With Moderately Severe to Severe Non-proliferative Diabetic Retinopathy
Brief Title: Non-proliferative Diabetic Retinopathy Treated With Runcaciguat
Acronym: NEON-NPDR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20739; 2020-002333-15 (EudraCT Number)
Record Dates: First submitted 2021-01-22; First posted 2021-01-25 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Retinopathy
Keywords: Non-proliferative Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — BAY 1101042

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-masked study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Runcaciguat (BAY1101042) (Experimental)
  Interventions: Drug: Runcaciguat (BAY1101042)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Runcaciguat (BAY1101042) — Oral dose of runcaciguat
  Arms: Runcaciguat (BAY1101042)
Other: Placebo — Oral dose of matching placebo
  Arms: Placebo

SUMMARY:
This Phase 2 study is conducted to investigate the safety and efficacy of runcaciguat in the treatment of diabetic retinopathy. To assess efficacy, the retinal morphology will be investigated by 7-field color fundus photography for central assessment of the diabetic retinopathy severity score, or DRSS. Two-step DRSS improvement at 24 weeks of treatment will be the primary efficacy endpoint. DRSS assessments are repeated after completion of 48 weeks of treatment. In addition, vision threatening complications will be recorded throughout the study and assessed as secondary efficacy endpoint.

ELIGIBILITY:
Main Inclusion Criteria:

* Moderately severe to severe NPDR in the study eye: Diabetic Retinopathy Severity Scale (DRSS) levels 47 or 53
* Diabetes type 1 or 2
* Best corrected visual acuity (BCVA) Early Treatment Diabetic Retinopathy Study (ETDRS) letter score in the study eye of ≥69 letters (approximate Snellen equivalent of 20/40 or better)

Main Exclusion Criteria:

* Presence or history of macular edema involving the center of the macula
* Any kind of neovascular growth in the study eye, including anterior segment neovascularization
* Arterial hypotension with systolic blood pressure < 100 or diastolic blood pressure < 60mmHg
* Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) above 3 x Upper limit of normal (ULN) or bilirubin ≥ 1.5 ULN at screening, known ascites
* Estimated glomerular filtration rate (eGFR CKD-EPI) below 30 ml/min/1.73 m^2 at screening
* Any prior systemic anti-Vascular endothelial growth factor (VEGF) treatment or IVT anti-VEGF treatment in the study eye
* Any prior intraocular steroid injection in the study eye
* Any prior grid or focal laser photocoagulation within 500 microns of the foveal center or any prior Pan-retinal photocoagulation (PRP) in the study eye
* Use of nitrates or Nitric oxide (NO) donors (such as amyl nitrate) in any form including topical; Phosphodiesterase 5 (PDE5) inhibitors, nonspecific PDE inhibitors within 1 week or less than 5 half-lives (whichever is longer) before first study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (55):
- United States (11):
  - Retinal Consultants Medical Group, Inc, Modesto, California
  - Florida Retina Consultants, Lakeland, Florida
  - Eye Associates of Pinellas, Pinellas Park, Florida
  - Cumberland Valley Retina Consultants | Hagerstown, MD, Hagerstown, Maryland
  - Mid Atlantic Retina Specialists - Hagerstown, Hagerstown, Maryland
  - Austin Research Center for Retina, Austin, Texas
  - Austin Retina Associates - Central, Austin, Texas
  - Retinal Consultants of Texas - Bellaire, Bellaire, Texas
  - Gulf Coast Eye Institute / Valley Retina Institute, McAllen, Texas
  - Retinal Consultants of Texas - San Antonio, San Antonio, Texas
  - Retina Consultants of Texas - The Woodlands, The Woodlands, Texas
- Bulgaria (5):
  - Eye center Sveti Luka, Plovdiv
  - UMHAT Sveti Georgi, Plovdiv
  - SEHAT Pentagram, Sofia
  - Diagnostic-Consultative Center Alexandrovska | Sofia, Bulgaria, Sofia
  - Sveta Petka Eye Hospital, Varna
- Czechia (4):
  - Ocni klinika Oftex, Pardubice
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Všeobecná fakultní nemocnice v Praze, Prague
  - Axon Clinical, s.r.o., Prague
- Denmark (5):
  - Aalborg Universitetshospital - Øjenafdelingen, Aalborg
  - Aarhus Universitetshospital, Aarhus N
  - Rigshospitalet Glostrup - Øjensygdomme, Glostrup Municipality
  - Odense Universitetshospital, Dept of Ophtalmology, Odense C
  - Sjællands Universitetshospital Roskilde - Hormon og stofskiftesygdomme, Roskilde
- NUVISAN GmbH Neu-Ulm, Neu-Ulm, Bavaria, Germany
- Riga East University Hospital, Bikernieki, Ophthalmology Clinic, Riga, Latvia
- Netherlands (3):
  - Academic Medical Center Dept Ophthalmology, Amsterdam
  - Universitair Medisch Centrum St. Radboud, Nijmegen
  - ETZ Elisabeth Ziekenhuis, Tilburg
- Poland (5):
  - Biokinetica S.A, Józefów
  - Klinika Okulistyczna "Jasne Blonia" Sp. z o.o, Lodz
  - Osrodek Chirurgii Oka prof. Zagorskiego Sp. z o.o., Rzeszów
  - Ind. Spec. Prakt. Lek. Dr W. Jedrzejewski, Tarnowskie Góry
  - NZOZ Centrum Badan Klinicznych, Wroclaw
- Portugal (4):
  - AIBILI, Coimbra
  - CHUC - Hospitais da U. Coimbra - Servico de Oftalmologia, Coimbra
  - Centro Hospitalar Universitario do Porto, Porto
  - Centro Hospitalar Universitario de Sao Joao | Polo Porto - Centro de Investigacao e Ensaios Clinicos, Porto
- Clinical Emergency County Hospital, Cluj-Napoca, Romania
- Slovakia (2):
  - Fakultna Nemocnica s poliklinikou F.D.Roosevelta, Banská Bystrica
  - Nemocnica Poprad, a.s., Poprad
- Spain (4):
  - Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario del Henares, Coslada, Madrid
  - Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen de la Macarena, Seville
- Switzerland (4):
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - Inselspital Universitätsspital Bern, Bern
  - University Eye Hospital Jules Gonin, Lausanne
  - Stadtspital Triemli, Zurich
- United Kingdom (5):
  - Gloucestershire Hospitals NHS Foundation Trust | Gloucestershire Royal Hospital - Gloucestershire Retinal Research Group, Gloucester, Gloucestershire
  - Sunderland Eye Infirmary, Sunderland, Tyne and Wear
  - Bristol Eye Hospital, Bristol
  - Moorfields Eye Hospital, London
  - King's College Hospital NHS Foundation Trust | King's College Hospital - Neurology Department, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 39 study centers in Europe and US that randomized 109 participants from 17 MAR 2021 (first patient first visit) to 22 APR 2024 (last patient last visit).
Pre-assignment Details: Out of the 224 screened participants, 109 participants were randomized and started treatment. 115 participants did not pass screening. The primary reason for screen failure was that one or more inclusion or exclusion criteria were not met by the participant.
Groups:
- Runcacigat (BAY1101042): Participants received runcaciguat gastrointestinal therapeutic system (GITS) tablets and were treated following an intra-individual dose-titration design with three titration steps.
- Placebo: Participants received matching placebo GITS tablets.
Period: Overall Study
Arm/Group | Runcacigat (BAY1101042) | Placebo
Started (randomized and assigned to treatment) | 56 | 53
Completed (All participants who completed the week 48 treatment) | 38 | 44
Not Completed | 18 | 9
Not completed — Adverse Event | 12 | 4
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal cirterion met | 2 | 2
Not completed — Other | 1 | 0
Not completed — Non-compliance | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included 109 participants (all randomized participants)
Groups:
- Total: Total of all reporting groups
Arm/Group | Runcacigat (BAY1101042) | Placebo | Total
Number analyzed (Participants) | 56 | 53 | 109
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.4 (12.7) | 57.9 (11.5) | 57.1 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 31 | 31 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 54 | 50 | 104
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Improvement in DRSS by ≥ 2 Steps at 48 Weeks of Treatment in the Study Eye
Description: DRSS (Diabetic Retinopathy Severity Scale) is measured on a 13-point scale and was graded centrally for the study.
Time Frame: At 48 weeks of treatment
Population: per protocol set: all full analysis set (FAS) participants of the respective study part without validity findings.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Runcacigat (BAY1101042) | Placebo
Number analyzed (Participants) | 51 | 52
percentage of participants | 0.0 [0.0 to 4.7] | 1.9 [0.2 to 8.7]
Statistical Analysis 1: Comparison: Runcacigat (BAY1101042) vs Placebo; Test type: Other — Bayesian inference with non-informative priors; Point estimate = -0.015, 95% CI 2-sided [-0.080 to 0.029] — Median of posterior distribution

2. Secondary Outcome: Percentage Participants With Vision Threatening Complications (VTC) at 48 Weeks of Treatment in the Study Eye
Description: VTC are defined as occurrence of any of the following AEs:
  * Proliferative diabetic retinopathy (PDR) (DRSS ≥61)
  * Any ocular neo-vascularization (retinal or anterior-segment neovascularization)
  * Center-involved (central Early Treatment Diabetic Retinopathy Study [ETDRS] subfield) DME
  * Drop of Best corrected visual acuity (BCVA) of 10 letters or more from baseline
Time Frame: At 48 weeks
Population: per protocol set: all full analysis set (FAS) participants of the respective study part without validity findings.
Measure: Number; unit: percentage of participants
Arm/Group | Runcacigat (BAY1101042) | Placebo
Number analyzed (Participants) | 51 | 52
percentage of participants | 17.6 | 11.5

3. Secondary Outcome: Percentage of Participants With ≥ 2 Steps Improvement in DRSS at 24 Weeks of Treatment in the Study Eye
Description: DRSS (Diabetic Retinopathy Severity Scale) is measured on a 13-point scale and was graded centrally for the study.
Time Frame: At 24 weeks of treatment
Population: per protocol set: all full analysis set (FAS) participants of the respective study part without validity findings.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Runcacigat (BAY1101042) | Placebo
Number analyzed (Participants) | 51 | 52
percentage of participants | 0.0 [0.0 to 4.8] | 0.0 [0.0 to 4.7]

4. Secondary Outcome: Percentage of Participants With ≥ 3 Steps Improvement in DRSS at 48 Weeks of Treatment on the for Persons Scale
Description: DRSS (Diabetic Retinopathy Severity Scale) is measured on a 13-point scale and was graded centrally for the study.
Time Frame: At 48 weeks of treatment
Population: per protocol set: all full analysis set (FAS) participants of the respective study part without validity findings.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Runcacigat (BAY1101042) | Placebo
Number analyzed (Participants) | 51 | 52
percentage of participants | 0.0 [0.0 to 4.7] | 1.9 [0.2 to 8.7]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Event (TEAE)
Time Frame: From first dosing up to 28 days after last dose of study intervention
Population: Safety analysis set (SAF): All participants of the respective study part who took at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Runcacigat (BAY1101042) | Placebo
Number analyzed (Participants) | 56 | 53
Participants | 53 | 44

6. Other Pre Specified Outcome: Percentage of Participants With < 3 Steps Deterioration in DRSS at 48 Weeks of Treatment on the for Persons Scale
Description: DRSS (Diabetic Retinopathy Severity Scale) is measured on a 13-point scale and was graded centrally for the study.
Time Frame: At 48 weeks of treatment
Population: per protocol set: all full analysis set (FAS) participants of the respective study part without validity findings.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Runcacigat (BAY1101042) | Placebo
Number analyzed (Participants) | 51 | 52
percentage of participants | 78.4 [65.8 to 88.0] | 80.8 [68.5 to 89.7]

ADVERSE EVENTS:
Time Frame: After the first study intervention up to 28 days after the end of study intervention, with an average up to 53 weeks. Adverse event reporting for the all-cause mortality considers all deaths that occurred at any time during the study before the last contact, with an average of/ up to 54 weeks.
Groups:
- Runcaciguat (BAY1101042): Participants received runcaciguat gastrointestinal therapeutic system (GITS) tablets and were treated following an intra-individual dose-titration design with three titration steps.
Arm/Group | Runcaciguat (BAY1101042) | Placebo
All-Cause Mortality (participants affected / at risk) | 2/56 | 0/53
Serious Adverse Events (participants affected / at risk) | 9/56 | 3/53
Other Adverse Events (participants affected / at risk) | 50/56 | 32/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Runcaciguat (BAY1101042) (N=56) | Placebo (N=53)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (2) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (2)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (2) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Runcaciguat (BAY1101042) (N=56) | Placebo (N=53)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Erythropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 2 (2) | 3 (4)
Diabetic retinopathy (Eye disorders) | 3 (3) | 2 (2)
Dry eye (Eye disorders) | 1 (1) | 3 (3)
Retinal exudates (Eye disorders) | 3 (3) | 0 (0)
Retinal haemorrhage (Eye disorders) | 3 (3) | 2 (2)
Vision blurred (Eye disorders) | 3 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (5) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 16 (28) | 10 (17)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 6 (7) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (5) | 5 (7)
Fatigue (General disorders) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Tooth infection (Infections and infestations) | 4 (4) | 1 (1)
COVID-19 (Infections and infestations) | 5 (5) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Blood creatinine increased (Investigations) | 4 (4) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 4 (4) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 6 (12) | 2 (6)
Headache (Nervous system disorders) | 6 (24) | 4 (4)
Depression (Psychiatric disorders) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 4 (4)
Hypotension (Vascular disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT04722991/Prot_002.pdf
  • Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT04722991/SAP_003.pdf